CLINICAL TRIAL: NCT06262087
Title: The Combined FIFA 11+ and Change of Direction Training on Knee Valgus Angle During Cutting in Male Soccer Players
Brief Title: The Combined FIFA 11+ and Change of Direction Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Komsak Sinsurin, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MU-CIRB 2023/044.2203
Record Dates: First submitted 2024-01-30; First posted 2024-02-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Rehabilitation; Physical Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIFA 11+ program combined with COD training (Experimental): Participants in an experimental group will perform the FIFA 11+ program combined with COD training.
  Interventions: Behavioral: Change of direction training; Behavioral: FIFA 11+ program
- FIFA 11+ (Active Comparator): Participants in the control group will perform the FIFA 11+ program.
  Interventions: Behavioral: FIFA 11+ program

INTERVENTIONS:
Behavioral: Change of direction training — The experimental group is implemented FIFA 11+ program combined with COD training
  Arms: FIFA 11+ program combined with COD training
Behavioral: FIFA 11+ program — The experimental group is implemented FIFA 11+ program.

SUMMARY:
The study has investigated the effects of adding change of direction (COD) training to the FIFA 11+ on lower extremity performance in soccer players. The investigators are interested in knee valgus angle during cutting which is typically suggested as a critical risk of anterior cruciate ligament injury. Peak knee valgus angle during cutting is expected to reduce immediately after adding COD training to the FIFA 11+.

ELIGIBILITY:
Inclusion Criteria:

* Soccer players

Exclusion Criteria:

* Having experience of serious injury such as, ACL injury and chronic ankle instability
* Having experience of lower limb surgery such as, bone fracture, tendon rupture, or ligament rupture
* Having current musculoskeletal injuries such as, muscle sprain
* Attending other prevention program or similar study especially on lower extremity
* Soccer player who are unable to perform level 3 of part 2 of the FIFA 11+ prevention program

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-06-07 (Actual); Study Completion 2025-12-07 (Actual)

PRIMARY OUTCOMES:
Peak knee valgus angle | At pre-training and immediate post-training of prevention program
  Knee valgus angle during cutting tests will be assessed before and after training for both groups. Two-dimensional analysis will be used to capture cutting movement and knee valgus angle will be extracted in the free software analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- FFC league in Cambodia, Phnom Penh, Phnom Penh, Cambodia

IPD SHARING:
Plan to Share IPD: Undecided
We will consider in the future.